CLINICAL TRIAL: NCT02151058
Title: Whitening Action of a Hydrogen Peroxide/Sodium Fluoride Containing Mouth Rinse: A 2 Week Randomized Controlled Trial
Brief Title: A Clinical Trial to Test the Effect of a Marketed Mouth Rinse on Stain Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CO-131219112750-CTOC
Record Dates: First submitted 2014-05-27; First posted 2014-05-30 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2014-10

CONDITIONS: Tooth Stain
Keywords: Staining; Intensity; Area
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Negative Control, 035000513007 (Other): Colgate® Regular Cavity Protection
  Interventions: Drug: Colgate® Regular Cavity Protection
- Experimental Mouth Rinse, 19545-118 (Experimental)
  Interventions: Drug: Experimental Mouth Rinse
- Active Comparator: Mouth Rinse 037000089872 (Active Comparator): Crest® 3D White Multi-Care Whitening Rinse, Glamorous White, Fresh Mint
  Interventions: Other: Crest® 3D White Multi-Care Whitening Rinse, Glamorous White, Fresh Mint

INTERVENTIONS:
Drug: Colgate® Regular Cavity Protection — Brushing twice daily with an ADA - Accepted fluoride - containing dentifrice (Colgate Cavity Protection)
  Arms: Negative Control, 035000513007
Drug: Experimental Mouth Rinse — Brushing twice daily with an ADA - Accepted containing toothpaste, followed by rinsing with 10 mL for 60 seconds with the investigational product.
  Arms: Experimental Mouth Rinse, 19545-118
Other: Crest® 3D White Multi-Care Whitening Rinse, Glamorous White, Fresh Mint — Brushing twice daily with an ADA - Accepted containing toothpaste, followed by rinsing with 15 mL for 60 seconds with the active comparator.
  Arms: Active Comparator: Mouth Rinse 037000089872

SUMMARY:
The whitening action of an investigative hydrogen peroxide/sodium fluoride containing mouth rinse will be evaluated through stain removal using mean Lobene Stain Index over 14 days compared to a currently marketed hydrogen peroxide containing whitening mouth rinse (Crest® 3D White Multi-Care Whitening Rinse, Glamorous White, Fresh Mint). A currently marketed toothpaste (Colgate® Cavity Protection) will be included as the negative control in order to compare to brushing alone.

225 healthy volunteers will be enrolled in this two week study. Volunteers who qualify to be in this study will have an equal chance of being assigned to one of the three treatment groups. Volunteers will have a total of 5 clinic visits including 1) screening, 2) baseline 3) Day 4 (after 3 days of use), Day 8 (after 7 days of use) and Day 15 (after 14 days of use). Volunteers will maintain a diary at home to record each treatment use. Examinations for oral hard/soft tissue assessment and extrinsic tooth stain after the subject brushes with water and floss will be completed at Baseline and repeated at Clinic Visits 3, 4, and 5, which are on Days 4, 8 and 15 post baseline (i.e., after 3, 7, and 14 days of product use).

DETAILED DESCRIPTION:
Approximately 225 generally healthy subjects that meet the required inclusion/exclusion criteria will be enrolled in this 2 week, examiner-blind, single center, randomized, controlled, parallel-group clinical trial to ensure that approximately 215 subjects complete the study. At baseline, the prescreened subjects will present to the clinical site for baseline examinations (oral tissue assessment, extrinsic tooth stain assessment). Subjects will brush with water, then floss, have an oral exam and tooth stain assessment. Subjects will be randomly assigned to one of three groups using a randomized code provided by the sponsor:

* Negative Control - Brushing twice daily with an ADA - Accepted fluoride-containing dentifrice (Colgate® Cavity Protection).
* Brushing twice daily with an ADA - Accepted fluoride-containing dentifrice (Colgate® Cavity Protection) followed by rinsing twice daily with 10 ml for 60 seconds with an investigative peroxide and fluoride containing mouth rinse
* Brushing twice daily with an ADA - Accepted fluoride-containing dentifrice (Colgate® Cavity Protection) followed by rinsing twice daily with 15 ml for 60 seconds with Crest® 3D White Multi-Care Whitening Rinse, Glamorous White, Fresh Mint

Immediately after randomization, subjects will begin use of their assigned test treatment. The site staff will supervise the first rinse treatment, and rinse treatments occurring on examination days. The negative control group will not have supervised brushing at the clinic to avoid the possibility of changing their usual brushing habits. All home use will be unsupervised and following label instructions. Subjects will be required to maintain a diary card to document twice-daily product use by recording their assigned oral care routine. For Clinic Visit 3, 4, and 5, subjects will be instructed to not use the treatment rinse in the morning prior to their clinic visit, because that treatment rinse will be supervised during their clinic visit. Subjects may brush as normal in the morning prior to these clinic visits.

During the study, subjects will follow their usual interdental cleaning (e.g. flossing) and dietary habits. Subjects will not be allowed to use any other unassigned oral care products (mouth rinse, dentifrice, or other tooth whitening products), or have their teeth professionally polished, bleached, or whitened by a dentist or hygienist.

Examinations for oral hard/soft tissue assessment and extrinsic tooth stain after the subject brushes with water and floss will be repeated at Clinic Visits 3, 4, and 5, which are on Days 4, 8 and 15 post baseline (i.e., after 3, 7, and 14 days of product use). Compliance will be evaluated at Visits 3, 4, and 5 by weighing residual volumes of returned mouth rinses and by reviewing the subject diary. Subjects will receive the ADA-Accepted fluoride containing dentifrice and a soft bristled toothbrush at their baseline visit.

During the course of the study, subjects may use an interdental cleaning device to remove impacted food between the teeth and may continue using an interdental cleaning device regularly if it is part of their usual oral care regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 65 years.
2. Able to comprehend and follow the requirements of the study (including availability on scheduled visit dates) based upon research site personnel's assessment;
3. Able to provide written informed consent;
4. Male or non-pregnant, non-lactating female (self-reported)
5. Male and female subjects with reproductive potential must agree to practice a medically acceptable form of birth control during the study and for 30 days following the last dose of investigational product
6. Medically acceptable forms of birth control that may be used by the subject and/or his/her partner
7. Able to read and understand the local language;
8. Able to follow study procedures;
9. Willing for this to be the only investigational product used during this time period; and
10. Willing and able to comply with all study procedures and attend the scheduled visits for the duration of the study.
11. Subject must have at least 2 natural anterior teeth, each having a mean Lobene composite score of ≥ 1.5 on the facial surfaces as assessed by the Investigator

Exclusion Criteria:

1. Suspected alcohol or substance abuse (e.g., amphetamines, benzodiazepines, cocaine, and marijuana) opiates.
2. Females who are pregnant or breastfeeding.
3. Males with a pregnant partner or a partner who is currently trying to become pregnant.
4. Known sensitivity or history of significant adverse effects to any of the investigational products.
5. Significant unstable or uncontrolled medical condition which may interfere with a subject's participation in the study.
6. Participated in tooth stain removal trials in the least 3 months
7. Participation in any other clinical study within 30 days of Visit 1.
8. Subjects who are related to those persons involved directly or indirectly with the conduct of this study (i.e., principal investigator, sub-investigators, study coordinators, other site personnel, employees of Johnson & Johnson subsidiaries, contractors of Johnson & Johnson, and the families of each).
9. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Milleman Milleman, DDS, MPA, Principal Investigator — Salus Research Inc.
Locations (1):
- Salus Research Inc, Fort Wayne, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Negative Control: Colgate® Regular Cavity Protection Toothpaste (Brushing Only)
- Crest 3D: Colgate® Regular Cavity Protection Toothpaste followed by Crest® 3D Whitening Rinse (Brushing followed by Mouth Rinse)
- Investigative Mouth Rinse: Colgate® Regular Cavity Protection Toothpaste followed by Investigative Hydrogen Peroxide/Sodium Fluoride Mouth Rinse (Brushing followed by Mouth Rinse)
Period: Overall Study
Arm/Group | Negative Control | Crest 3D | Investigative Mouth Rinse
Started | 45 | 91 | 91
Completed | 43 | 90 | 86
Not Completed | 2 | 1 | 5
Not completed — Withdrawal by Subject | 1 | 1 | 3
Not completed — Lost to Follow-up | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Negative Control | Crest 3D | Investigative Mouth Rinse | Total
Number analyzed (Participants) | 45 | 91 | 91 | 227
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (12.57) | 43.3 (12.15) | 44.0 (12.40) | 43.8 (12.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 60 | 69 | 164
  Male | 10 | 31 | 22 | 63
Region of Enrollment [Number; unit: participants]
  USA | 45 | 91 | 91 | 227

OUTCOME MEASURES:

1. Primary Outcome: Lobene Stain Index Composite Score at Day 15
Description: Tooth stain surface and stain intensity were assessed by using scores on the Lobene Stain Index (two part visual scale), scored 0 - 3. Where 0 = no stain, 1 = light stain, 2 = moderate stain and 3 = heavy stain. The second part of the scale examined the surface of the tooth on a scale of 0-3, where 0= no stain, 1 = covering up to 1/3 of the region, 2 = covering > 1/3 to 2/3 of the region and 3 = covering > 2/3 of the region.
  The mean composite score (0-9) was determined by multiplying the individual tooth stain surface and stain intensity scores and summing then dividing by the number of regions scored for the subject (or tooth).
Time Frame: 15 Days
Population: Analysis was based on the Full Analysis Set, which included all randomized subjects who used study product and had baseline and at least one post-baseline efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Negative Control | Crest 3D | Investigative Mouth Rinse
Number analyzed (Participants) | 43 | 90 | 86
units on a scale | 2.568 (0.0821) | 1.909 (0.0568) | 1.575 (0.0580)
Statistical Analysis 1: Comparison: Negative Control vs Crest 3D; The null hypothesis was no difference in mean outcome between treatment groups. The alternative hypothesis was a difference in mean outcome between treatment groups; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.659, 95% CI 2-sided [-0.8559 to -0.4622], Standard Error of Mean 0.0999
Statistical Analysis 2: Comparison: Negative Control vs Investigative Mouth Rinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided). Hypotheses were tested according to a hierarchical strategy; Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.993, 95% CI 2-sided [-1.1909 to -0.7946], Standard Error of Mean 0.1005
Statistical Analysis 3: Comparison: Crest 3D vs Investigative Mouth Rinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided). Hypotheses were tested according to a hierarchical strategy; Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.334, 95% CI 2-sided [-0.4937 to -0.1737], Standard Error of Mean 0.0812

2. Secondary Outcome: Lobene Stain Index Composite Score at Day 4
Description: as for outcome 1
Time Frame: 4 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Negative Control | Crest 3D | Investigative Mouth Rinse
Number analyzed (Participants) | 43 | 90 | 88
units on a scale | 2.527 (0.0665) | 2.242 (0.0459) | 2.200 (0.0464)
Statistical Analysis 1: Comparison: Negative Control vs Crest 3D; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.286, 95% CI 2-sided [-0.4450 to -0.1263], Standard Error of Mean 0.0809
Statistical Analysis 2: Comparison: Negative Control vs Investigative Mouth Rinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.328, 95% CI 2-sided [-0.4877 to -0.1679], Standard Error of Mean 0.0811
Statistical Analysis 3: Comparison: Crest 3D vs Investigative Mouth Rinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.520, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.042, 95% CI 2-sided [-0.1709 to 0.0866], Standard Error of Mean 0.0653

3. Secondary Outcome: Lobene Stain Index Composite Score at Day 8
Description: as for outcome 1
Time Frame: 8 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Negative Control | Crest 3D | Investigative Mouth Rinse
Number analyzed (Participants) | 43 | 90 | 87
units on a scale | 2.536 (0.0798) | 2.023 (0.0551) | 1.852 (0.0561)
Statistical Analysis 1: Comparison: Negative Control vs Crest 3D; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.513, 95% CI 2-sided [-0.7043 to -0.3217], Standard Error of Mean 0.0971
Statistical Analysis 2: Comparison: Negative Control vs Investigative Mouth Rinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.685, 95% CI 2-sided [-0.8770 to -0.4925], Standard Error of Mean 0.0975
Statistical Analysis 3: Comparison: Crest 3D vs Investigative Mouth Rinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.030, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.172, 95% CI 2-sided [-0.3268 to -0.0168], Standard Error of Mean 0.0786

4. Secondary Outcome: Lobene Stain Index Area Scores at Day 4
Description: Tooth stain surface was assessed by using scores on the Lobene Stain Index scored 0 - 3, where 0= no stain, 1 = covering up to 1/3 of the region, 2 = covering > 1/3 to 2/3 of the region, and 3 = covering > 2/3 of the region.
Time Frame: 4 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Negative Control | Crest 3D | Investigative Mouth Rinse
Number analyzed (Participants) | 43 | 90 | 88
units on a scale | 1.621 (0.0304) | 1.538 (0.0209) | 1.502 (0.0212)
Statistical Analysis 1: Comparison: Negative Control vs Crest 3D; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.026, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.083, 95% CI 2-sided [-0.1556 to -0.0102], Standard Error of Mean 0.0369
Statistical Analysis 2: Comparison: Negative Control vs Investigative Mouth Rinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.002, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.118, 95% CI 2-sided [-0.1917 to -0.0451], Standard Error of Mean 0.0372
Statistical Analysis 3: Comparison: Crest 3D vs Investigative Mouth Rinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.234, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.035, 95% CI 2-sided [-0.0940 to 0.0231], Standard Error of Mean 0.0297

5. Secondary Outcome: Lobene Stain Index Area Scores at Day 8
Description: as for outcome 4
Time Frame: 8 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Negative Control | Crest 3D | Investigative Mouth Rinse
Number analyzed (Participants) | 43 | 90 | 87
units on a scale | 1.615 (0.0468) | 1.439 (0.0321) | 1.265 (0.0327)
Statistical Analysis 1: Comparison: Negative Control vs Crest 3D; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.002, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.176, 95% CI 2-sided [-0.2882 to -0.0644], Standard Error of Mean 0.0568
Statistical Analysis 2: Comparison: Negative Control vs Investigative Mouth Rinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.351, 95% CI 2-sided [-0.4638 to -0.2378], Standard Error of Mean 0.0573
Statistical Analysis 3: Comparison: Crest 3D vs Investigative Mouth Rinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.174, 95% CI 2-sided [-0.2648 to -0.0841], Standard Error of Mean 0.0458

6. Secondary Outcome: Lobene Stain Index Area Scores at Day 15
Description: as for outcome 4
Time Frame: 15 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Negative Control | Crest 3D | Investigative Mouth Rinse
Number analyzed (Participants) | 43 | 90 | 86
units on a scale | 1.629 (0.0520) | 1.382 (0.0357) | 1.131 (0.0366)
Statistical Analysis 1: Comparison: Negative Control vs Crest 3D; Treatment and baseline value as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.247, 95% CI 2-sided [-0.3713 to -0.1226], Standard Error of Mean 0.0631
Statistical Analysis 2: Comparison: Negative Control vs Investigative Mouth Rinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.498, 95% CI 2-sided [-0.6236 to -0.3722], Standard Error of Mean 0.0638
Statistical Analysis 3: Comparison: Crest 3D vs Investigative Mouth Rinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.251, 95% CI 2-sided [-0.3516 to -0.1503], Standard Error of Mean 0.0511

7. Secondary Outcome: Lobene Stain Index Intensity Scores at Day 4
Description: Tooth stain surface was assessed by using scores on the Lobene Stain Index scored 0 - 3, where 0= no stain, 1 = light stain, 2 = moderate stain, and 3 = heavy stain.
Time Frame: 4 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Negative Control | Crest 3D | Investigative Mouth Rinse
Number analyzed (Participants) | 43 | 90 | 88
units on a scale | 1.651 (0.0306) | 1.527 (0.0211) | 1.483 (0.0214)
Statistical Analysis 1: Comparison: Negative Control vs Crest 3D; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.124, 95% CI 2-sided [-0.1970 to -0.0504], Standard Error of Mean 0.0372
Statistical Analysis 2: Comparison: Negative Control vs Investigative Mouth Rinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.168, 95% CI 2-sided [-0.2413 to -0.0941], Standard Error of Mean 0.0373
Statistical Analysis 3: Comparison: Crest 3D vs Investigative Mouth Rinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.145, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.044, 95% CI 2-sided [-0.1034 to 0.0152], Standard Error of Mean 0.0301

8. Secondary Outcome: Lobene Stain Index Intensity Scores at Day 8
Description: as for outcome 7
Time Frame: 8 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Negative Control | Crest 3D | Investigative Mouth Rinse
Number analyzed (Participants) | 43 | 90 | 87
units on a scale | 1.668 (0.0409) | 1.438 (0.0283) | 1.355 (0.0288)
Statistical Analysis 1: Comparison: Negative Control vs Crest 3D; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.230, 95% CI 2-sided [-0.3282 to -0.1321], Standard Error of Mean 0.0497
Statistical Analysis 2: Comparison: Negative Control vs Investigative Mouth Rinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.313, 95% CI 2-sided [-0.4113 to -0.2141], Standard Error of Mean 0.0500
Statistical Analysis 3: Comparison: Crest 3D vs Investigative Mouth Rinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.042, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.083, 95% CI 2-sided [-0.1621 to -0.0031], Standard Error of Mean 0.0404

9. Secondary Outcome: Lobene Stain Index Intensity Scores at Day 15
Description: as for outcome 7
Time Frame: 15 Days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Negative Control | Crest 3D | Investigative Mouth Rinse
Number analyzed (Participants) | 43 | 90 | 86
units on a scale | 1.671 (0.0447) | 1.396 (0.0309) | 1.206 (0.0316)
Statistical Analysis 1: Comparison: Negative Control vs Crest 3D; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.275, 95% CI 2-sided [-0.3820 to -0.1679], Standard Error of Mean 0.0543
Statistical Analysis 2: Comparison: Negative Control vs Investigative Mouth Rinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.464, 95% CI 2-sided [-0.5724 to -0.3565], Standard Error of Mean 0.0548
Statistical Analysis 3: Comparison: Crest 3D vs Investigative Mouth Rinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided); Treatment and baseline value as covariates; Mean Difference (Final Values) = -0.190, 95% CI 2-sided [-0.2767 to -0.1023], Standard Error of Mean 0.0442

ADVERSE EVENTS:
Time Frame: Day 15 ± 2 days, +30 days for serious adverse events.
Description: Adverse events were systematically collected at each study visit through Visit 5 (Day 15 ± 2 days). Serious adverse events were reported through 30 days after product use. Spontaneously reported adverse events collected outside of the regularly scheduled visits were also recorded.
Arm/Group | Negative Control | Crest 3D | Investigative Mouth Rinse
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/91 | 0/91
Other Adverse Events (participants affected / at risk) | 0/45 | 0/91 | 0/91

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigator agreed not to publish the study results without prior sponsor approval.